CLINICAL TRIAL: NCT05621434
Title: Inetetamab, Pyrotinib and Chemotherapy in Combination for First-line Treatment of HER2-positive Recurrent/Metastatic Breast Cancer
Brief Title: A Study to Evaluate Inetetamab + Pyrotinib + Chemotherapy in Previously Untreated HER2-Positive Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Fan Wu, Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K2022-025-01
Record Dates: First submitted 2022-11-09; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: HER2-positive Recurrent/Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Drug Therapy; Injections

STUDY DESIGN:
Intervention Model Description: single arm study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inetetamab, pyrotinib, chemotherapy (Experimental): Inetetamab: was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  pyrotinib: 400 mg once daily orally within 30 minutes after a meal at the same time each day.
  chemotherapy:Taxanes (paclitaxel, docetaxel, liposomal paclitaxel, nabpaclitaxel), vinorelbine, capecitabine, eribulin, and other chemotherapeutic agents indicated in advanced breast cancer are permitted. Refer to the appropriate package insert for dosage and administration recommendations.
  Interventions: Drug: Inetetamab, pyrotinib, chemotherapy

INTERVENTIONS:
Drug: Inetetamab, pyrotinib, chemotherapy — Inetetamab: was administered as an intravenous (IV) loading dose of 8mg/kg q3w on Day 1 of Cycle 1 (1 Cycle length = 21 days), and 6mg/kg q3w on Day 1 of subsequent cycles, until investigator-assessed radiographic or clinical progressive disease, unmanageable toxicity, or study termination.
  pyrotinib: 400 mg once daily orally within 30 minutes after a meal at the same time each day.
  chemotherapy:Taxanes (paclitaxel, docetaxel, liposomal paclitaxel, nabpaclitaxel), vinorelbine, capecitabine, eribulin, and other chemotherapeutic agents indicated in advanced breast cancer are permitted. Refer to the appropriate package insert for dosage and administration recommendations.
  Other Names: Inetetamab for injection; Pyrotinib maleate

SUMMARY:
Studies H0648g and M77001 confirmed that the combination of trastuzumab with taxanes significantly improved TTP and OS, establishing the status of trastuzumab combined with taxanes as first-line standard therapy.The CLEOPATRA and PUFFIN studies confirmed that trastuzumab combined with pertuzumab achieved PFS of 18.7 and 16.5 months, respectively, and became today 's first-line standard regimen for advanced HER2 + breast cancer. Pyrotinib acts on the intracellular segment of HER2 receptor and can inhibit tumor cell growth by covalently binding to the ATP binding site in the intracellular tyrosine kinase region and blocking the activation of downstream signaling pathways. The mechanism of action of the macromolecular drug trastuzumab combined with the small molecular drug pyrotinib dual-target in the treatment of HER2-positive breast cancer is complementary and has a synergistic anti-tumor effect. In 2022, the ESMO conference reported the results of a phase III trial of pyrotinib combined with trastuzumab combined with docetaxel in advanced HER2-positive breast cancer with an LBA, with the primary endpoint of investigator-assessed PFS.The results showed a significant 59% reduction in the risk of disease progression or death compared with 10.4 months in the trastuzumab plus docetaxel arm and 24.3 months in the pyrotinib arm.

Inetetamab is a monoclonal antibody against the IV domain of the HER2 receptor with the same Fab segment as trastuzumab and different amino acid sequences from trastuzumab at positions 359 and 361 of the Fc segment heavy chain constant region, Antibody-dependent cell-mediated cytotoxicity (ADCC) was 1.11-fold higher than trastuzumab. PFS reached 11.1 months in the first-line subgroup analysis of the Phase III registration study of Inetetamab (HOPES study), which was similar to historical data from trastuzumab first-line treatment of HER2-positive metastatic breast cancer, with comparable safety. The results of this study contribute to further understanding the efficacy and safety of first-line treatment with Inetetamab Combined with Pyrotinib and Chemotherapy in HER2-positive recurrent/metastatic breast cancer patients.

DETAILED DESCRIPTION:
This Prospective, multicenter study will include 63 patients with first-line patients with HER2-positive recurrent/metastatic breast cancer. After providing written informed consent, patients receiving Inetetamab in combination with pyrotinib and investigator 's choice chemotherapy. The effectiveness of the combined treatment will be evaluated by MRI every two treatment cycles. If the disease progresses, the participant will withdraw from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 ~ 75 years old, female;
2. Patients with HER2-positive breast cancer defined as immunohistochemical (IHC) test + + +, or FISH test positive;
3. According to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, at least one measurable lesion exists;
4. ECOG PS score 0-1 points;
5. No systemic antitumor therapy (except first line endocrine therapy) in relapse/metastasis;
6. If prior anti-HER2 therapy (including trastuzumab, trastuzumab biosimilar, Inetetamab, pertuzumab, tyrosine kinase inhibitors such as pyrotinib, T-DM1) was used in the (neo) adjuvant phase, the interval between the end of anti-HER2 therapy to the diagnosis of relapse/metastasis was ≥ 12 months;
7. Adequate organ function;
8. Expected survival ≥ 3 months;
9. Patients voluntarily sign informed consent, have good compliance and are willing to cooperate in follow-up.

Exclusion Criteria:

1. Known to have a history of hypersensitivity to the drug components of this protocol;
2. Investigators judged that they were not suitable for systemic chemotherapy;
3. Endocrine therapy drugs were used within 14 days before baseline;
4. Active brain metastases;
5. Only bone or skin as target lesions;
6. Patients with other malignant tumors within 5 years, excluding cured cervical carcinoma in situ, cutaneous basal cell carcinoma or squamous cell carcinoma;
7. Grade≥3 peripheral neuropathy according to CTCAE 5.0 criteria;
8. Patients who have previously received more than the following cumulative doses of anthracyclines: doxorubicin or liposomal doxorubicin > 360 mg/m2, epirubicin > 720 mg/m2, mitoxantrone > 120 mg/m2, others (such as other anthracyclines or multiple anthracyclines, cumulative dose > 360 mg/m2 of doxorubicin);
9. Received major surgical procedures or significant trauma within 4 weeks before randomization, or patients are expected to receive major surgical treatment;
10. Serious heart problems or discomfort;
11. Dysphagia, chronic diarrhea, intestinal obstruction and other factors affecting administration and absorption;
12. History of immunodeficiency, including HIV infection, or suffering from other acquired, congenital immunodeficiency diseases, or history of organ transplantation; 13. Participated in other drug clinical studies within 4 weeks before screening;

14. Presence of third space effusion (such as pleural effusion and ascites) that cannot be controlled by drainage or other methods; 15. Pregnant or lactating female patients, women of childbearing age who cannot take effective contraceptive measures throughout the trial; 16. With severe concomitant diseases or interfere with the planned treatment or any other condition that is not suitable for participating in this study, such as active hepatitis B, lung infection requiring treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2022-12-10 (Estimated); Primary Completion 2024-12-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Tumor assessments every 6 weeks from randomization to radiographical PD or death from any cause, whichever occurred first，up to the primary completion date (up to 2 years)
  PFS was defined as the time from first dose to first documented radiographical progressive disease (PD) using RECIST version 1.1, or death from any cause , whichever occurred first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Tumor assessments every 6 weeks from Baseline until radiographical progressive disease (PD), death (whichever occurred first), up to the primary completion date (up to 2 years)
  An objective response was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) determined by investigator using RECIST v1.1 on two consecutive occasions ≥4 weeks apart
Clinical Benefit Rate (CBR) | Tumor assessments every 6 weeks from Baseline until radiographical progressive disease (PD), death (whichever occurred first), up to the primary completion date (up to 2 years)
  Clinical benefit rate was defined as the percentage of participants with confirmed best overall response of complete response (CR) or partial response (PR) or stable disease（SD）>6 months determined by investigator using RECIST v1.1 on two consecutive occasions ≥4 weeks apart.
Number of Adverse Events using NCI CTCAE 5.0 [Safety and Tolerability] | From signing the informed consent to 30 days after last dose
  Number of Adverse Events using NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jian Liu, PHD, Principal Investigator — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will indicate whether Inetetamab Combined with Pyrotinib and Chemotherapy treatment of HER2-Positive Recurrent/Metastatic Breast Cancer is safe and effective
Supporting Information: Study Protocol
Time Frame: 6 months to 5 years after publication
Access Criteria: Unlimited